CLINICAL TRIAL: NCT03311997
Title: The Proximal Hamstring Avulsion Clinical Trial - Nonoperative Treatment Compared With Suture Anchor Reinsertion of Proximal Hamstrings Avulsions
Brief Title: The Proximal Hamstring Avulsion Clinical Trial - Operative or Nonoperative Treatment
Acronym: PHACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Linkoeping University (Other Government); Lund University (Other); Örebro University, Sweden (Other); Umeå University (Other); Karolinska Institutet (Other); University of Oslo (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UU2017/170
Record Dates: First submitted 2017-10-10; First posted 2017-10-17 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Hamstring Tendon Injury
Keywords: RCT; Hamstring; Suture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Personell assessing functional performance of patients are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-operative treatment (No Intervention): Active rehabilitation program
- Operative treatment (Active Comparator): Surgical reattachment of hamstring tendons using suture anchors followed by active rehabilitation program
  Interventions: Procedure: Surgical reattachment of hamstring tendons

INTERVENTIONS:
Procedure: Surgical reattachment of hamstring tendons — operatively reattachment of the tendons using suture anchor
  Arms: Operative treatment

SUMMARY:
The purpose of this study is to provide reliable evidence on how to best treat proximal hamstrings avulsions, and our primary aim is to compare the reported outcome of patients treated non-operatively with patients treated with suture anchor reattachment of the tendons using the Perth Hamstrings Assessment Tool (PHAT) at 24 months.

DETAILED DESCRIPTION:
The treatment of proximal hamstrings avulsions is controversial and patients with this injury will get treatment recommendations based not on scientific evidence but on personal preferences of their surgeon. The literature is totally devoid of studies comparing the two treatment options; non-operative and operative treatment. In Sweden, it is probably more common to treat these injuries nonoperatively. This is in contrast to existing literature that suggests that better outcomes are expected with operative treatment. However, there is a very clear publication bias in the literature. In fact, of the more than 40 published clinical studies, only a handful mentions the results of non-operatively treated injuries.

In a systematic review examining 13 original studies, patient satisfaction ranged from 88% to 100% after surgical treatment. In nine of the studies strength of hamstrings were reported and ranged from 78% to 101% of the uninjured side. However, residual pain is common, ranging from 8 to 61% in a group of 203 patients and in a recent unpublished study the lower extremity functional score were similar in patients treated by either modality. Additionally, serious nerve injuries after surgery have been reported and infection, anchor failure and re-rupture occur. The reoperation rate in a study by Sarimo et al. was 12%.

This study is a prospective, multicentre, preference-tolerant, randomized controlled, non-inferiority trial comparing operative to non-operative treatment of proximal hamstrings avulsions. The study will include a concurrent prospective observational cohort.

The eligible study population will consist of patients with an acute, avulsion of hamstrings tendons diagnosed in a hospital in Sweden, or Norway and subsequently referred to one of the study sites. All patients fulfilling the inclusion and not meeting the exclusion criteria will be asked to participate in the study. After the patient´s enrolment has been confirmed and informed consent is obtained a set of questionnaires is provided for background data on medical history, activity levels and a recall assessment of the pre-injury functional status. When these questionnaires are completed, the patient is randomized.

If the patient is randomized to non-operative treatment an appointment with a physiotherapist follows and the study rehabilitation protocol is explained. If the patient is randomized to surgery, the procedure is scheduled at the earliest convenient time but no later than 2 weeks from inclusion. The surgical procedure and rehabilitation protocol is standardized among sites. The same rehabilitation protocol is used for both treatment groups.

Participation in this study will last 24 months. In-person participant follow-up visits will occur at enrollment (baseline), at-surgery, 3 months, 6 months, 12 months and 24 months post-surgery. Data for outcomes will be collected at follow-up visit and a MRI will be performed at 24 months.

ELIGIBILITY:
Inclusion criteria

* age of the patient at injury between 30 and 70
* MRI shows a complete avulsion of at least two of three tendons from the insertion at the ischial tubercule
* physical examination supports the diagnosis; e.g. a positive hip extension test, palpable defect and/or local tenderness and hematoma
* patient has a moderate to high activity level
* patient has linguistic and mental ability to understands study program explained in Swedish, Finnish, Norwegian or English
* time from injury to inclusion in study is less than 4 weeks

A patient with moderate to high activity level is defined as any patient that is ambulatory in the community and participates in some type of strenuous activity at work or in spare time on a regular basis. Any patient that skis, goes for an occasional run, takes long walks in the woods, climbs ladders or physically manages a large garden have an activity level that is at least moderate.

Exclusion criteria

* diabetes with secondary complications
* previous major lower extremity injury or disease with sequelae
* moderate or severe liver, pulmonary, kidney, psychiatric or heart disease that significantly increases the risk for complications after operative treatment
* severe obesity (BMI>35)
* alcohol or drug abuse
* high energy injury or combinations of injuries affecting the lower extremity

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Perth Hamstrings Assessment Tool (PHAT) | 24 months post inclusion
  The PHAT is a 8-item instrument that measures pain, function and discomfort of the hamstrings. Primary endpoint at 24 months (measured at 3, 6, 12, and 24 months). The maximum score is 100 indicating no symptoms and high function.

SECONDARY OUTCOMES:
Lower extremity functional scale (LEFS) | 24 months post inclusion
  LEFS is a 30-item instrument that measure patient perceived function of the lower extremities. Primary endpoint at 24 months (measured at 3, 6, 12, and 24 months). The maximum possible score is 80 points, indicating very high function.
Maximal isokinetic strength of hamstrings | 24 months post inclusion
  The difference between the two treatment groups in the mean ratio between the injured and uninjured side of the maximum isokinetic force during knee flexion and hip extension measured by a dynamometer. Primary endpoint at 24 months (measured at 3, 6, 12, and 24 months).
Timed step test | 24 months post inclusion
  The difference between the two treatment groups in the mean ratio between the injured and uninjured side of the functional timed step test. Primary endpoint at 24 months (measured at 3, 6, 12, and 24 months).
Single hop test | 24 months post inclusion
  The difference between the two treatment groups in the mean ratio between the injured and uninjured side of the single leg hop test. Primary endpoint at 24 months (measured at 3, 6, 12, and 24 months).
Hamstrings muscle volume and density | 24 months post inclusion
  Volume and density measured by DIXON MRI at 24 months

OTHER OUTCOMES:
Adverse events | up until last follow-up at 24 months
  Peripheral neurological injury and symptoms, infection, wound complications, thromboembolic disease and any serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Jonsson, MD., Ph.D, Principal Investigator — Uppsala University
Locations (10):
- Norway (2):
  - Bergen University Hospital, Bergen
  - Oslo University Hospital, Oslo
- Sweden (8):
  - Linköping University Hospital, Linköping
  - Malmö University Hospital, Malmo
  - Örebro University Hospital, Örebro
  - Östersund Hospital, Östersund
  - Södersjukhuset, Stockholm
  - Danderyd hospital, Stockholm
  - Norrlands University Hospital, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 6 months of study completion
Access Criteria: Data access request will be reviewed by independent University leaders. Requestors will be required to sign DAA

REFERENCES:
- [Background] Iyer VG. Iatrogenic injury to the sciatic nerve during surgical repair of proximal hamstring avulsion. Muscle Nerve. 2015 Sep;52(3):465-6. doi: 10.1002/mus.24678. Epub 2015 May 14. No abstract available. PMID 25847226
- [Background] Blakeney WG, Zilko SR, Edmonston SJ, Schupp NE, Annear PT. Proximal hamstring tendon avulsion surgery: evaluation of the Perth Hamstring Assessment Tool. Knee Surg Sports Traumatol Arthrosc. 2017 Jun;25(6):1936-1942. doi: 10.1007/s00167-016-4214-y. Epub 2016 Jun 25. PMID 27344550
- [Background] Harris JD, Griesser MJ, Best TM, Ellis TJ. Treatment of proximal hamstring ruptures - a systematic review. Int J Sports Med. 2011 Jul;32(7):490-5. doi: 10.1055/s-0031-1273753. Epub 2011 May 11. PMID 21563032
- [Background] Barry MJ, Palmer WE, Petruska AJ. A Proximal Hamstring Injury--Getting Off a Slippery Slope. JAMA Intern Med. 2016 Jan;176(1):15-6. doi: 10.1001/jamainternmed.2015.6795. No abstract available. PMID 26618607
- [Background] Mehta SP, Fulton A, Quach C, Thistle M, Toledo C, Evans NA. Measurement Properties of the Lower Extremity Functional Scale: A Systematic Review. J Orthop Sports Phys Ther. 2016 Mar;46(3):200-16. doi: 10.2519/jospt.2016.6165. Epub 2016 Jan 26. PMID 26813750
- [Background] Sarimo J, Lempainen L, Mattila K, Orava S. Complete proximal hamstring avulsions: a series of 41 patients with operative treatment. Am J Sports Med. 2008 Jun;36(6):1110-5. doi: 10.1177/0363546508314427. Epub 2008 Mar 4. PMID 18319349
- [Background] van der Made AD, Reurink G, Gouttebarge V, Tol JL, Kerkhoffs GM. Outcome After Surgical Repair of Proximal Hamstring Avulsions: A Systematic Review. Am J Sports Med. 2015 Nov;43(11):2841-51. doi: 10.1177/0363546514555327. Epub 2014 Nov 10. PMID 25384502
- [Derived] Pihl E, Laszlo S, Rosenlund AM, Kristoffersen MH, Schilcher J, Hedbeck CJ, Skorpil M, Micoli C, Eklund M, Skoldenberg O, Frihagen F, Jonsson KB. Operative versus Nonoperative Treatment of Proximal Hamstring Avulsions. NEJM Evid. 2024 Aug;3(8):EVIDoa2400056. doi: 10.1056/EVIDoa2400056. Epub 2024 Jul 18. PMID 39023393
- [Derived] Pihl E, Kristoffersen MH, Rosenlund AM, Laszlo S, Berglof M, Ribom E, Eriksson K, Frihagen F, Mattila VM, Schilcher J, Eklund M, Snellman G, Skorpil M, Skoldenberg O, Hedbeck CJ, Jonsson K. The proximal hamstring avulsion clinical trial (PHACT)-a randomised controlled non-inferiority trial of operative versus non-operative treatment of proximal hamstrings avulsions: study protocol. BMJ Open. 2019 Sep 13;9(9):e031607. doi: 10.1136/bmjopen-2019-031607. PMID 31519683

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT03311997/SAP_000.pdf